CLINICAL TRIAL: NCT03081962
Title: Effect of Intraperitoneal Irrigation With Antibiotic Solution, Triclosan-impregnated Sutures for Fascial Closure and Mupirocin Ointment Over the Skin Staples, on Surgical-site Infection After Laparoscopic Colorectal Surgery
Brief Title: Effect of a Combination of Bundles on Surgical-site Infection After Elective Colorectal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Principal Investigator, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HGUE-2016-23
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The election of the intervention will be performed following a randomization model. Only the care provider will know the assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bundle application (Experimental): The patients in this group will undergo an intraperitoneal irrigation with clindamycin and gentamicin solution, fascial closure with triclosan impregnated sutures and application of Mupirocin ointment over the skin staples
  Interventions: Drug: Bundle; Procedure: Standard care
- Standard care (Active Comparator): The patients in this group will follow a standard care, including decontamination of the skin during surgery with chlorhexidine alcohol solution, administration of systemic antibiotic prophylaxis and application of thermal blanket to avoid hypothermia. In the standard care, the fascial closure will be performed with a polyglactin suture (without Triclosan impregnation).
  Interventions: Procedure: Standard care

INTERVENTIONS:
Drug: Bundle — Combination of antibiotic intraperitoneal irrigation with gentamicin and clindamycin solution, use of Triclosan-impregnated sutures and mupirocin application over the skin staples.
  Other Names: Combination of 3 measures for SSI prevention
  Arms: Bundle application
Procedure: Standard care — Standard care measures include decontamination of the skin during surgery with chlorhexidine alcohol solution, administration of systemic antibiotic prophylaxis and application of thermal blanket to avoid hypothermia. In the standard care protocol, the fascial closure will be performed with a polyglactin suture (without Triclosan impregnation).
  Other Names: Standard care measures for SSI prevention

SUMMARY:
A prospective randomized clinical trial will be performed. Patients will be randomized in 2 groups. The experimental group will undergo the combined application of intraperitoneal irrigation with clindamycin and gentamicin solution, fascial closure with Triclosan-impregnated sutures and application of mupirocin ointment over the skin staples, in addition to the standard care measures. The control group undergo only the standard care measures.

Incisional surgical-site infection will be investigated.

DETAILED DESCRIPTION:
A prospective randomized clinical trial will be performed. Patients will be randomized in 2 groups. The experimental group will undergo the combined application of intraperitoneal irrigation with clindamycin (600mg) and gentamicin (240 mg) solution in 250 ml of normal saline, fascial closure with Triclosan-impregnated polyglactin suture and application of mupirocin ointment over the skin staples, in addition to the standard care measures. The control group undergo only the standard care measures, including decontamination of the skin during surgery with chlorhexidine alcohol solution, administration of systemic antibiotic prophylaxis and application of thermal blanket to avoid hypothermia. In the control group, the fascial closure will be performed with a polyglactin suture (without Triclosan impregnation).

Incisional surgical-site infection will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer undergoing elective laparoscopic colorectal surgery with curative aims.

Exclusion Criteria:

* Chronic renal failure
* Immunodeficiency status, including uncontrolled Type 2 diabetes mellitus and patients under corticoid or immunosuppresive treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Incisional surgical site infection | 30 days postoperatively
  Incisional surgical site infection will be evaluated up to the 30th postoperative day by an epidemiology nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Llavero, Study Director — Hospital General Elche
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ruiz-Tovar J, Llavero C, Morales V, Gamallo C. Effect of the application of a bundle of three measures (intraperitoneal lavage with antibiotic solution, fascial closure with Triclosan-coated sutures and Mupirocin ointment application on the skin staples) on the surgical site infection after elective laparoscopic colorectal cancer surgery. Surg Endosc. 2018 Aug;32(8):3495-3501. doi: 10.1007/s00464-018-6069-4. Epub 2018 Jan 18. PMID 29349539